CLINICAL TRIAL: NCT03202043
Title: Sensitivity of Skin Carotenoid Status to Detect Changes in Intake of Varying Levels of Vegetables
Brief Title: The Juice Study: Sensitivity of Skin Carotenoid Status to Detect Change in Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GFHNRC150
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight | interventions — Fruit and Vegetable Juices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High dose vegetable juice (Experimental): Subject will consume high dose vegetable juice daily for 8 weeks.
  Interventions: Other: High dose vegetable juice
- Medium dose vegetable juice (Experimental): Subject will consume medium dose vegetable juice daily for 8 weeks.
  Interventions: Other: Medium dose vegetable juice
- Low dose vegetable juice (Experimental): Subject will consume low dose vegetable juice daily for 8 weeks.
  Interventions: Other: Low dose vegetable juice
- Control bottled water (Other): Subject will consume control bottled water daily for 8 weeks.
  Interventions: Other: Control bottled water

INTERVENTIONS:
Other: High dose vegetable juice — High dose (13 fl oz) vegetable juice
  Arms: High dose vegetable juice
Other: Medium dose vegetable juice — Medium dose (10 fl oz) vegetable juice
  Arms: Medium dose vegetable juice
Other: Low dose vegetable juice — Low dose (5.5 fl oz) vegetable juice
  Arms: Low dose vegetable juice
Other: Control bottled water — Control (12 fl oz) bottled water
  Arms: Control bottled water

SUMMARY:
This study is designed to see if drinking a tomato-based vegetable juice will increase skin carotenoids.

DETAILED DESCRIPTION:
The US Dietary Guidelines for Americans recommends that individuals consume approximately 2-4 c of vegetables each day to reduce risk of chronic disease, but current methods for assessing intake are either inaccurate (self-report) or invasive (blood carotenoid levels). Recent research indicates that skin carotenoid status may be a useful biomarker of vegetable intake, but the sensitivity to dose in unknown. In this study, we propose to test the dose-response of skin carotenoids to consumption of 3 different levels of vegetable juice (with a control group receiving water). We will test skin carotenoids in two ways: using resonance Raman spectroscopy (RRS), which we have previously validated, and with a new technique, pressure mediated reflection spectroscopy (RS; the "Veggie Meter"). We will compare the two techniques during an 8-week provided tomato-based juice intervention. Skin carotenoid readings will be compared to blood carotenoid concentrations and single nucleotide polymorphisms (SNPs) of genes related to the uptake, transport, and metabolism of carotenoids will be examined in blood and saliva.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5-29.9 kg/m2

Exclusion Criteria:

* weigh less than 110 lbs
* currently dieting to lose weight
* allergic to tomatoes or vegetables
* pregnant, lactating, or planning to become pregnant
* currently use tobacco products or vape
* eat more that 2 cups of vegetables per day
* have high blood sugar (≥200 mg/dL)
* have high blood pressure (≥140/90 mm Hg)
* have a medical condition such as diabetes or high blood pressure
* taking medication that lowers cholesterol or triglycerides

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2019-05-21 (Actual)

PRIMARY OUTCOMES:
Change in skin carotenoid concentration as measured by pressure-mediated reflection spectroscopy (RS) | 0, 4, 8 weeks
  Pressure-mediated reflection spectroscopy (RS) is used to measure tissue carotenoids. RS intensity can be used as a measure for total carotenoid content in the measured tissue volume.

SECONDARY OUTCOMES:
Usual intake of carotenoid-rich foods and beverages | 0,4,8 weeks
  A 44-item food frequency questionnaire of the top carotenoid-rich foods and beverages will be developed to measure carotenoid intake from a person's usual diet.

CONTACTS AND LOCATIONS:
Overall Officials: James Roemmich, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Norman AC, Palmer DG, Moran NE, Roemmich JN, Casperson SL. Association of Candidate Single-Nucleotide Polymorphism Genotypes With Plasma and Skin Carotenoid Concentrations in Adults Provided a Lycopene-Rich Juice. J Nutr. 2024 Jul;154(7):1985-1993. doi: 10.1016/j.tjnut.2024.05.022. Epub 2024 May 24. PMID 38797482
- [Derived] Casperson SL, Roemmich JN, Larson KJ, Hess JM, Palmer DG, Jahns L. Sensitivity of Pressure-Mediated Reflection Spectroscopy to Detect Changes in Skin Carotenoids in Adults Without Obesity in Response to Increased Carotenoid Intake: A Randomized Controlled Trial. J Nutr. 2023 Feb;153(2):588-597. doi: 10.1016/j.tjnut.2023.01.002. Epub 2023 Jan 6. PMID 36894250
- See also: Grand Forks Human Nutrition Research Center Current Nutrition Studies — https://www.ars.usda.gov/plains-area/gfnd/gfhnrc/docs/nutrition-studies/nutrition-studies/

DOCUMENTS (1):
  • Informed Consent Form (2019-04-05): https://cdn.clinicaltrials.gov/large-docs/43/NCT03202043/ICF_000.pdf